CLINICAL TRIAL: NCT02587728
Title: Collection of Peripheral Blood Samples From Patients With Carpal Tunnel Syndrome for Laboratory Screening of Amyloidosis
Brief Title: Carpal Tunnel/Amyloidosis Blood Sample Study
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, James Hoffman, MD, Associate Professor of Clinical, University of Miami
Other Study IDs: 20140503
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Carpal Tunnel Syndrome; Amyloidosis
MeSH Terms: conditions — Carpal Tunnel Syndrome; Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genome DNA extracted peripheral blood mononuclear cells (PBMCs)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carpal Tunnel Blood Draw: Participants with confirmed diagnosis of Carpal Tunnel Syndrome who will undergo blood draw for laboratory analysis for amyloidosis.

SUMMARY:
Carpal tunnel is an early manifestation of amyloidosis in a significant minority of patients. This specimen collection protocol will allow the investigators to screen patients with carpal tunnel syndrome for amyloidosis.

DETAILED DESCRIPTION:
The investigators propose to assess a high risk population of patients, those with carpal tunnel syndrome, and systematically assess them for Amyloid Light-chain (AL) amyloidosis and Transthyretin-Related Amyloidosis (ATTR) with simple laboratory blood tests. The combination of serum immunofixation electrophoresis together with serum free light chain (FLC) assay approaches 100% sensitivity for identifying the monoclonal protein underlying the illness in patients with AL amyloidosis. In addition to this, testing for transthyretin gene mutations will allow the investigators to identify patients with ATTR. The investigators believe this simple screening panel (serum immunofixation and serum FLC assay and transthyretin mutation analysis) may allow the investigators to identify patients early in the course of their disease, at which point the investigators can intervene with effective treatment and spare patients a significant amount of morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with diagnosed carpal tunnel syndrome based on Electromyography (EMG) results.
* 2. Patients with electrographic confirmation of median neuropathy at the wrist
* 3. Age ≥18 years
* 4. Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* 1. Patients receiving hemodialysis
* 2. Known amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients within 24 months of confirmed diagnosis of Carpal Tunnel Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2016-02-24 (Actual); Primary Completion 2017-02-07 (Actual); Study Completion 2017-02-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants Identified with Amyloidosis | Up to 5 years
  Number of carpal tunnel syndrome patients identified with amyloidosis, which will be stratified into mild, moderate or severe

CONTACTS AND LOCATIONS:
Overall Officials: James Hoffman, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No